CLINICAL TRIAL: NCT00915954
Title: Growth Hormone Feedback In Patients With Acromegaly, Type 2 Diabetes Mellitus, And Healthy Adults
Brief Title: Growth Hormone Feedback to Insulin-like Growth Factor-I (IGF-1) and Oral Glucose Tolerance Test (OGTT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Odelia Cooper, Staff Physician II, Cedars-Sinai Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 17015
Record Dates: First submitted 2009-06-05; First posted 2009-06-08 (Estimated); Results first posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Acromegaly; Type 2 Diabetes Mellitus
Keywords: Acromegaly; Type 2 diabetes mellitus; recombinant human Insulin like growth factor 1 (IGF1); oral glucose tolerance test
MeSH Terms: conditions — Acromegaly; Diabetes Mellitus, Type 2 | interventions — Glucose Tolerance Test

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Active Acromegaly (Active Comparator): Placebo, oral glucose tolerance test, and subcutaneous administration of recombinant human IGF-1 will be given at visits 2, 3, and 4 respectively. All visits will be performed within a 4 week period.
  Interventions: Diagnostic Test: Oral Glucose Tolerance Test; Diagnostic Test: Subcutaneous administration of recombinant human IGF-1; Diagnostic Test: Placebo
- Type 2 Diabetes Mellitus(DM) (Active Comparator): Placebo, oral glucose tolerance test, and subcutaneous administration of recombinant human IGF-1 will be given at visits 2, 3, and 4 respectively. All visits will be performed within a 4 week period.
  Interventions: Diagnostic Test: Oral Glucose Tolerance Test; Diagnostic Test: Subcutaneous administration of recombinant human IGF-1; Diagnostic Test: Placebo
- Heathy Controls (Active Comparator): Placebo, oral glucose tolerance test, and subcutaneous administration of recombinant human IGF-1 will be given at visits 2, 3, and 4 respectively. All visits will be performed within a 4 week period.
  Interventions: Diagnostic Test: Oral Glucose Tolerance Test; Diagnostic Test: Subcutaneous administration of recombinant human IGF-1; Diagnostic Test: Placebo

INTERVENTIONS:
Diagnostic Test: Oral Glucose Tolerance Test — Participants will have their blood drawn for a baseline value and then will be asked to drink a beverage with 75 grams of sugar. Blood will then be drawn every 30 minutes for 2 hours.
Diagnostic Test: Subcutaneous administration of recombinant human IGF-1 — Participants will receive a subcutaneous injection of recombinant human IGF-1 followed by a series of blood draws.
Diagnostic Test: Placebo — Participants will receive a subcutaneous injection of saline followed by a series of blood draws.

SUMMARY:
Growth hormone (GH) and Insulin-like growth factor-I (IGF-I) secretion are altered in acromegaly and type 2 Diabetes Mellitis (DM). The secretion of GH is mediated by central hypothalamic hormones (GH Releasing Hormone and somatostatin) as well as peripheral factors providing feedback inhibition (IGF-I and glucose, among others). The purpose of this study is to compare growth hormone suppression after an oral glucose tolerance test (OGTT) to growth hormone suppression after recombinant human IGF-I (rhIGF-I) administration. This study will recruit participants with active acromegaly, type 2 diabetes mellitus, and healthy control subjects. Each participant will undergo a screening evaluation, and three subsequent visits. Each participant will receive a placebo subcutaneous injection, OGTT, and administration of rhIGF-I, on separate visit days. Glucose, insulin, GH, bioactive IGF-I and IGF-I binding proteins will be measured after each intervention. Results will be compared between the three groups. It is predicted that the administration of rhIGF-I will demonstrate GH suppression in all healthy subjects and subjects with type 2DM. Some acromegaly subjects may demonstrate GH suppression in response to IGF-I administration, but not to the degree seen in healthy subjects or type 2 DM. OGTT will demonstrate suppression of GH in normal subjects, and will show attenuated suppression in type 2 DM and a failure of suppression in acromegaly.

DETAILED DESCRIPTION:
Acromegaly is characterized by unrestrained growth hormone (GH) secretion and subsequent elevated insulin-like growth factor (IGF)-1 resulting from a benign somatotroph GH-secreting adenoma in the pituitary. In healthy individuals, the negative feedback loop regulating GH secretion is modulated in part by IGF-1, which inhibits basal GH secretion as well as GH secretion mediated by hypothalamic growth hormone releasing hormone (GHRH). IGF-1 also suppresses basal and GHRH-induced gene transcription and downregulates GH receptors in the periphery to limit local GH action. In acromegaly, somatotroph proliferation and transformation may lead to disrupted GH feedback regulation, leading to tonically elevated GH and IGF-1 levels that remain unrestrained.

Elevated serum IGF-1 levels in patients with acral or soft tissue overgrowth and/or disease-associated comorbidities is suggestive of the disorder, and demonstrated evidence of GH excess is required to confirm the diagnosis. The standard confirmatory diagnostic test for acromegaly is the oral glucose tolerance test (OGTT). In healthy adults, acute oral glucose administration suppresses GH secretion for 1-3 hours before rebounding; failure to suppress GH in response to a 75 g glucose load on OGTT indicates abnormal GH hypersecretion and thus confirms the acromegaly diagnosis.

This diagnostic approach, however, assumes that GH suppression after a glucose load is unaffected by factors other than acromegaly. Low GH levels have been reported in younger women after OGTT, and high GH levels are observed in those with anorexia nervosa, bulimia, and nutritional deficiencies. Whether and how these factors might affect OGTT interpretation in the diagnosis of acromegaly is unknown.

Importantly, poorly controlled diabetes mellitus also results in GH hypersecretion that may not suppress on OGTT. As an estimated one-quarter of patients with newly diagnosed acromegaly have impaired fasting glycemia or glucose intolerance, and one-quarter have frank diabetes, disruptions in the glucose/GH axis could undermine use of OGTT as a diagnostic tool. Earlier consensus recommendations cautioned against the use of OGTT in patients with impaired glucose metabolism; current recommendations do not advise this, although the risk of inducing hyperglycemia in these patients remains a concern.

Following on the investigators' earlier work describing the molecular basis for IGF-1 regulation of GH synthesis and its role in the negative feedback loop regulating GH secretion and action, the investigators considered whether recombinant human (rh) IGF-1 could reproducibly discriminate between normal and excessive GH secretion, and whether administering this peptide could be useful as an alternative to OGTT as a confirmatory diagnostic test for acromegaly.

In healthy subjects with an intact GH/IGF-1 feedback loop, rhIGF-1 administration markedly increases levels of circulating IGF-1 and suppresses GH, primarily by inhibiting hypothalamic-mediated GH secretion and blunting GH pulse amplitude, although effects on GH may be dose-dependent. rhIGF-1 administration in patients with obesity and diabetes has also been shown to suppress GH. By contrast, in patients with acromegaly, where the GH/IGF-1 feedback loop is usually not intact, rhIGF-1 administration fails to suppress, or attenuates, GH secretion and reduces exogenous GHRH responses while only minimally affecting GH pulsatility patterns .

Building on these observations, the investigators propose to analyze GH responses to rhIGF-1 administration and OGTT in non-acromegaly patients with type 2 diabetes mellitus (T2DM), nondiabetic patients with acromegaly, and healthy controls. The aims are to determine whether rhIGF-1 administration could be used to elicit a sufficiently distinct GH response in acromegaly versus those without acromegaly, without conferring adverse glycemic effects.

ELIGIBILITY:
Inclusion Criteria:

* Active acromegaly due to excess GH produced by a pituitary adenoma.
* Patients must have an elevated IGF-I compared to age and gender matched controls (as supplied by the laboratory) and fail to suppress GH to below 1 ng/ml after a standard 75g oral glucose tolerance test.
* Type 2 diabetes mellitus, defined by elevated fasting glucose ≥ 126 mg/dl (verified by two historical measurements), or plasma glucose ≥ 200 mg/dl two hours after a 75 g oral glucose load, or a random glucose ≥ 200 mg/dl.

Exclusion Criteria:

1. Acromegaly Group

   * Current medical therapy for acromegaly including dopamine agonists, somatostatin analogues, or growth hormone antagonists.
   * For subjects on current therapy the following washout periods may be used:

     * Cabergoline: 4 weeks
     * Bromocriptine: 1 week
     * Sandostatin LAR: 3 months
     * Short-acting octreotide: 1 week
     * Lanreotide: 3 months
     * Pegvisomant: 4 weeks
   * Subjects with a history of surgical therapy for treatment of acromegaly must have verification of active disease with verified elevated IGF-I for the subjects' age and gender compared to healthy controls (as supplied by the laboratory) (two measures) as well as a failure to suppress GH to below 1 ng/ml after OGTT.
   * Current treatment for insulin resistance or type 2 DM including oral or injection medications.
   * Fasting glucose ≥ 126 mg/dl at screening evaluation.
   * Evidence of hepatic or renal disease defined as elevated transaminases, elevated serum creatinine.
   * Pregnancy or breast feeding.
2. Type 2 diabetes mellitus group

   * Patients taking non-insulin medications for diabetes treatment will be excluded.
   * Diagnosis of acromegaly.
   * Evidence of hepatic or renal disease defined as elevated transaminases, elevated serum creatinine.
   * Pregnancy or breast feeding.
3. Healthy Control Group

   * History of diabetes mellitus or impaired glucose tolerance, history of acromegaly.
   * Fasting glucose ≥ 126 mg/dl at screening evaluation.
   * Evidence of hepatic or renal disease defined as elevated transaminases, elevated serum creatinine.
   * Pregnancy or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-12; Primary Completion 2013-08 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Odelia Cooper, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center Pituitary Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Heathly Controls: Placebo, oral glucose tolerance test, and subcutaneous administration of recombinant human IGF-1 will be given at visits 2, 3, and 4 respectively. All visits will be performed within a 4 week period.
  Oral Glucose Tolerance Test: Participants will have their blood drawn for a baseline value and then will be asked to drink a beverage with 75 grams of sugar. Blood will then be drawn every 30 minutes for 2 hours.
  Subcutaneous administration of recombinant human IGF-1: Participants will receive a subcutaneous injection of recombinant human IGF-1 followed by a series of blood draws.
  Placebo: Participants will receive a subcutaneous injection of saline followed by a series of blood draws.
Period: Overall Study
Arm/Group | Active Acromegaly | Type 2 Diabetes Mellitus(DM) | Heathly Controls
Started | 10 | 8 | 10
Completed | 10 | 8 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Acromegaly | Type 2 Diabetes Mellitus(DM) | Heathly Controls | Total
Number analyzed (Participants) | 10 | 8 | 10 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 6 | 8 | 22
  >=65 years | 2 | 2 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (18) | 54 (9) | 38 (17) | 46 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 5 | 12
  Male | 6 | 5 | 5 | 16
Region of Enrollment [Number; unit: participants]
  United States | 10 | 8 | 10 | 28

OUTCOME MEASURES:

1. Primary Outcome: Percentage With Growth Hormone (GH) Suppression to < 0.4 ng/ml
Description: Subjects underwent recombinant insulin like growth factor 1 (rhIGF1) suppression testing and growth hormone levels were measured at time 0, 15, 30, 60, 90, 120, and 180 minutes after injection of rhIGF-1. A response </= 0.4 ng/ml is considered a normal response in the healthy control and diabetic control subjects. The percentage of subjects with a normal GH suppression to </= 0.4 ng/ml was calculated.
Time Frame: Before injection and at time 15, 30, 60, 90, 120 and 180 minutes after rhIGF-1 injection on week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Active Acromegaly | Type 2 Diabetes Mellitus(DM) | Heathly Controls
Number analyzed (Participants) | 10 | 8 | 10
Participants | 0 | 7 | 8

2. Secondary Outcome: Median Insulin Like Growth Factor Binding Protein 1 (IGFBP-1) Area Under the Curve in Response to Placebo, Oral Glucose Tolerance Test (OGTT), and rhIGF1 Suppression Testing
Description: IGFBP1 levels were measured at time 0 prior to the injection and measured at 15, 30, 60, 90, 120, and 180 minutes after injection. The area under the curve of IGFBP1 was calculated for each subject and the medians calculated for each cohort during the placebo, OGTT, and rhIGF1 tests.
Time Frame: Before injection at time 0 and then at 15, 30, 60, 90, 120, and 180 minutes after injection for week 2, 3, and 4 for each cohort for placebo, OGTT, and rhIGF1, respectively.
Measure: Median (Full Range); unit: ng*min/mL
Arm/Group | Active Acromegaly | Type 2 Diabetes Mellitus(DM) | Heathly Controls
Number analyzed (Participants) | 10 | 8 | 10
ng*min/mL
  Placebo | 10927 [2963 to 85103] | 5079 [2317 to 12915] | 9105 [2645 to 16808]
  OGTT | 5603 [3758 to 63248] | 2538 [2207 to 28208] | 4266 [637 to 27870]
  IGF-1 suppression test | 10901 [3098 to 62873] | 7347 [1578 to 10911] | 7681 [3318 to 16256]

3. Secondary Outcome: Median Insulin Level in Response to Placebo, OGTT, and rhIGF1 Testing
Description: Insulin levels were measured at time 120 minutes after injection. Median insulin was calculated for each cohort during the placebo, OGTT, and rhIGF1 tests.
Time Frame: Measured at 120 minutes after injection for week 2, 3, and 4 for each cohort for placebo, OGTT, and rhIGF1, respectively.
Measure: Median (Full Range); unit: mU/L
Arm/Group | Active Acromegaly | Type 2 Diabetes Mellitus(DM) | Heathly Controls
Number analyzed (Participants) | 10 | 8 | 10
mU/L
  Placebo | 7 [3 to 16] | 9 [4 to 91] | 4 [0.5 to 6]
  OGTT | 55 [6 to 395] | 39.5 [22 to 217] | 41.5 [11 to 124]
  IGF-1 suppression test | 4 [0.5 to 13] | 4.5 [2 to 108] | 2.5 [0.5 to 9]

4. Secondary Outcome: Median Bioactive IGF-1 Area Under the Curve in Response to Placebo, OGTT, and rhIGF1 Testing
Description: Bioactive IGF-1 levels were measured at time 0 prior to the injection and measured at 15, 30, 60, 90, 120, and 180 minutes after injection. The area under the curve of bioactive IGF-1 was calculated for each subject and the medians calculated for each cohort during the placebo, OGTT, and rhIGF1 tests.
Time Frame: as for outcome 2
Measure: Median (Full Range); unit: ng*min/mL
Arm/Group | Active Acromegaly | Type 2 Diabetes Mellitus(DM) | Heathly Controls
Number analyzed (Participants) | 10 | 8 | 10
ng*min/mL
  Placebo | 716 [353 to 1154] | 291 [127 to 842] | 302 [138 to 902]
  OGTT | 699 [379 to 1038] | 270 [219 to 422] | 339 [89 to 874]
  IGF-1 suppression test | 1004 [853 to 1464] | 659 [108 to 876] | 642 [338 to 970]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the 4 weeks of the study period.
Arm/Group | Active Acromegaly | Type 2 Diabetes Mellitus(DM) | Heathly Controls
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 2/10 | 0/8 | 0/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Acromegaly (N=10) | Type 2 Diabetes Mellitus(DM) (N=8) | Heathly Controls (N=10)
Low blood pressure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — 4 hours after administration of glucola, the patient's blood pressure was checked prior to discharge from visit and was found to be low (85/42). Manual blood pressure was performed and was higher (95/47). Patient was asymptomatic throughout.
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — After receiving an injection of rhIGF-1, the participant developed a mild skin reaction that was present on the back and upper extremities. By the end of the study visit, the flushing and redness had gradually subsided.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes